CLINICAL TRIAL: NCT06190340
Title: A Phase 1, Single-center, Double-blind, Placebo-controlled Study to Evaluate Pharmacokinetics (PK) and Preliminary Efficacy of Multiple Oral Administrations of TNP-2092 Capsules in Healthy Subjects With Helicobacter Pylori Infection
Brief Title: A Phase 1 Study to Evaluate PK Profile of Multiple Oral Administrations of TNP-2092 Capsules in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TenNor Therapeutics (Suzhou) Limited (Industry)
Collaborators: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Organization: TenNor Therapeutics Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: TNP-2092-03
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — TNP-2092

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TNP-2092 capsules 100 mg (Experimental): Subjects received TNP-2092 capsules orally twice daily at the dose of 100 mg in the fed state for consecutive 14 days and received the last dose in the fed state on the morning of Day 15
  Interventions: Drug: TNP-2092 capsules
- TNP-2092 capsules 300 mg (Experimental): Subjects received TNP-2092 capsules orally twice daily at the dose of 300 mg in the fed state for consecutive 14 days and received the last dose in the fed state on the morning of Day 15
  Interventions: Drug: TNP-2092 capsules
- TNP-2092 capsules 600 mg (Experimental): Subjects received TNP-2092 capsules orally twice daily at the dose of 600 mg in the fed state for consecutive 14 days and received the last dose in the fed state on the morning of Day 15
  Interventions: Drug: TNP-2092 capsules
- Placebo (Placebo Comparator): Subjects received TNP-2092 placebo capsules orally twice daily in the fed state for consecutive 14 days and received the last dose in the fed state on the morning of Day 15
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TNP-2092 capsules — Administration orally.
  Other Names: Rifaquizinone capsules
  Arms: TNP-2092 capsules 100 mg; TNP-2092 capsules 300 mg; TNP-2092 capsules 600 mg
Drug: Placebo — Administration orally.
  Other Names: TNP-2092 placebo capsules
  Arms: Placebo

SUMMARY:
This study was a single-center, randomized, double-blind, placebo-controlled, dose-ascending multiple-dose-administration study. The aim of this study was to evaluate the safety, tolerability, and pharmacokinetic profile of TNP-2092 Capsules in asymptomatic healthy subjects with Helicobacter pylori infection, and to explore the preliminary efficacy of TNP-2092 Capsules in eradicating Helicobacter pylori.

DETAILED DESCRIPTION:
This study was a single-center, randomized, double-blind, placebo-controlled, dose-ascending multiple-dose-administration study. The aim of this study was to evaluate the safety, tolerability, and pharmacokinetic profile of TNP-2092 Capsules in asymptomatic healthy subjects with Helicobacter pylori infection, and to explore the preliminary efficacy of TNP-2092 Capsules in eradicating Helicobacter pylori.

In this study, three dose groups of 100 mg, 300 mg and 600 mg will be set up. The drug will be taken twice a day for 14 consecutive days, and last dose on the morning of Day 15. Fifteen subjects in each of the 100 mg and 300 mg dose groups will be randomized at a ratio of 4:1, with 12 subjects receiving the investigational product and 3 receiving placebo. Ten subjects in the 600 mg dose group will be randomized at a ratio of 4:1, with 8 subjects receiving the investigational product and 2 subjects receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

* Those who are fully informed of and understand this study and have signed the Informed Consent Form.
* Those who are willing to follow and able to complete all the trial procedures.
* Female subjects of childbearing potential must agree to abstinence or take effective contraceptive measures during the trial and at least 70 days (10 weeks) after administration.
* Male subjects must agree to abstinence or use condoms as a contraceptive measure during the trial and at least 70 days (10 weeks) after administration.
* Sex: male or female.
* Age: 18-45 years, including 18 and 45 years.
* BMI: 19.0-26.0 kg/m2, including 19.0 and 26.0 kg/m2.
* Those who do not smoke, or have smoked less than 5 cigarettes per day within 3 months before screening; those who do not drink alcohol, or have drunk less than 14 units of alcohol per week (1 unit of alcohol = 360 mL of beer or 45 mL of spirits with 40% alcohol content or 150 mL of wine) within 6 months before screening; those who have not smoked or drunk alcohol within 48 hours before admission to the study site.
* Subjects whose clinical laboratory test results are within the normal range or whose test results are abnormal but judged by the investigator to be of no clinical insignificance.
* Those with a positive 14C urea breath test (UBT) result.

Exclusion Criteria:

* Those with an allergic constitution, a history of allergic diseases or a history of drug allergy.
* Those with a history of alcohol or drug abuse in the past 10 years.
* Those who have donated blood within 3 months before enrollment.
* Those with regular use of any prescription/over-the-counter drugs, including vitamins, minerals, nutritional supplements or herbs, within 2 weeks before enrollment and during the study period.
* Those who have taken any drug that changes the activity of liver enzymes 28 days before taking the investigational product or during the study.
* Those who have participated in any clinical trials within 3 months before enrollment.
* Those with a history of eradication of Helicobacter pylori.
* Those who are suffering or have suffered from digestive tract diseases, including digestive tract ulcer, etc.
* Those with symptoms or past medical history of cardiovascular, respiratory, urinary, neurological, blood, immune, endocrine system diseases or tumor, mental illness, or any situation which, in the opinion of the investigator, may threaten the safety of the subjects or affect the correctness of the trial results.
* Those whose blood pressure remains above 140/90 mmHg after retest.
* Pregnant or lactating women.
* Those who are HIV positive, syphilis positive, hepatitis B surface antigen positive, hepatitis C antibody positive.
* Those who have had beverages or foods containing methylxanthine (coffee, tea, coke, chocolate, and energy drinks), grapefruit (fruit juice) and alcohol within 48 hours (2 days) before the clinical study.
* Other circumstances deemed by the investigator to be unsuitable for the subject to participate in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2017-09-26 (Actual); Study Completion 2017-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, MD, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TNP-2092 Capsules 100 mg | TNP-2092 Capsules 300 mg | TNP-2092 Capsules 600 mg | Placebo
Started | 12 | 12 | 8 | 8
Completed | 12 | 12 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Subjects received Placebo orally twice daily in the fed state for consecutive 14 days and received the last dose in the fed state on the morning of Day 15.
- Total: Total of all reporting groups
Arm/Group | TNP-2092 Capsules 100 mg | TNP-2092 Capsules 300 mg | TNP-2092 Capsules 600 mg | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 8 | 8 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 8 | 8 | 40
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (7.99) | 32.7 (7.75) | 33.5 (5.78) | 34.0 (6.70) | 32.1 (7.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 2 | 13
  Male | 9 | 8 | 4 | 6 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 12 | 12 | 8 | 8 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Positive rates of carbon 14 urea breath test (14C UBT) [Count of Participants; unit: Participants] | 12 | 12 | 8 | 8 | 40

OUTCOME MEASURES:

1. Primary Outcome: Safety of TNP-2092 by Assessment of the Number of Adverse Events (AEs)
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment.
Time Frame: Day 1 to Day 49
Population: All subjects who have received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | TNP-2092 Capsules 100 mg | TNP-2092 Capsules 300 mg | TNP-2092 Capsules 600 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 8 | 8
participants | 6 | 9 | 4 | 3

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve Over a Dosing Interval (AUC0-tau) on Day 1
Description: Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma Pharmacokinetics (PK) parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Time Frame: Day 1：Before administration (within 60 minutes), 0.5, 1, 2, 3, 4, 6, 8, 10 and 12 hours after administration
Population: All subjects who have been randomized into groups, have received at least one dose of study drug, and have at least one evaluable pharmacokinetic parameter.
Measure: Mean (Standard Deviation); unit: h*µg/L
Arm/Group | TNP-2092 Capsules 100 mg | TNP-2092 Capsules 300 mg | TNP-2092 Capsules 600 mg
Number analyzed (Participants) | 12 | 12 | 8
h*µg/L | 62.8 (34.4) | 190 (86.5) | 618 (310)

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of TNP-2092 on Day 1
Description: as for outcome 2
Time Frame: Day 1：Before administration (within 60 minutes), 0.5, 1, 2, 3, 4, 6, 8, 10 and 12 hours after administration
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | TNP-2092 Capsules 100 mg | TNP-2092 Capsules 300 mg | TNP-2092 Capsules 600 mg
Number analyzed (Participants) | 12 | 12 | 8
µg/L | 17.7 (8.38) | 46.4 (21.7) | 149 (78.4)

4. Primary Outcome: Time to Reach the Maximum Observed Plasma Concentration (Tmax) on Day 1
Description: as for outcome 2
Time Frame: Day 1：Before administration (within 60 minutes), 0.5, 1, 2, 3, 4, 6, 8, 10 and 12 hours after administration
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | TNP-2092 Capsules 100 mg | TNP-2092 Capsules 300 mg | TNP-2092 Capsules 600 mg
Number analyzed (Participants) | 12 | 12 | 8
h | 4 (1) | 4 (1) | 4 (0.8)

5. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve Extrapolated to Infinity (AUC0-inf) on Day 15
Description: as for outcome 2
Time Frame: Day 15: Before administration (within 60 minutes), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours after administration
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*µg/L
Arm/Group | TNP-2092 Capsules 100 mg | TNP-2092 Capsules 300 mg | TNP-2092 Capsules 600 mg
Number analyzed (Participants) | 12 | 12 | 8
h*µg/L | 96.5 (46.5) | 274 (114) | 701 (274)

6. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From the First Administration to the Last Measurable Plasma Concentration (AUC0-last) on Day 15
Description: as for outcome 2
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*µg/L
Arm/Group | TNP-2092 Capsules 100 mg | TNP-2092 Capsules 300 mg | TNP-2092 Capsules 600 mg
Number analyzed (Participants) | 12 | 12 | 8
h*µg/L | 93.3 (46.1) | 267 (112) | 692 (272)

7. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve Over a Dosing Interval (AUC0-tau) on Day 15
Description: Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma PK parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*µg/L
Arm/Group | TNP-2092 Capsules 100 mg | TNP-2092 Capsules 300 mg | TNP-2092 Capsules 600 mg
Number analyzed (Participants) | 12 | 12 | 8
h*µg/L | 90.7 (41.1) | 250 (105) | 657 (257)

8. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of TNP-2092 on Day 15
Description: as for outcome 2
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | TNP-2092 Capsules 100 mg | TNP-2092 Capsules 300 mg | TNP-2092 Capsules 600 mg
Number analyzed (Participants) | 12 | 12 | 8
µg/L | 21.7 (9.35) | 59.9 (30.2) | 167 (75.6)

9. Primary Outcome: Time to Reach the Maximum Observed Plasma Concentration (Tmax) Day 15
Description: as for outcome 2
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | TNP-2092 Capsules 100 mg | TNP-2092 Capsules 300 mg | TNP-2092 Capsules 600 mg
Number analyzed (Participants) | 12 | 12 | 8
h | 4 (0.9) | 3 (2) | 4 (0.5)

10. Primary Outcome: Half Life (t1/2) of TNP-2092 on Day 15
Description: as for outcome 2
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | TNP-2092 Capsules 100 mg | TNP-2092 Capsules 300 mg | TNP-2092 Capsules 600 mg
Number analyzed (Participants) | 12 | 12 | 8
h | 3.26 (1.29) | 7.3 (4.91) | 6.67 (2.57)

11. Primary Outcome: Number of Participants With Negative Results of 14 Urea Breath Test (14C UBT) at 4 to 6 Weeks After Last Dose
Description: Participants received 14 urea breath test [14C UBT] at 4 to 6 weeks after last dose.
Time Frame: Four to 6 weeks after the last dose of the study drugs.
Population: All the subjects who were randomized into groups
Measure: Number; unit: participants
Arm/Group | TNP-2092 Capsules 100 mg | TNP-2092 Capsules 300 mg | TNP-2092 Capsules 600 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 8 | 8
participants | 1 | 1 | 0 | 1

12. Primary Outcome: Accumulation Index Rac (AUC) of TNP-2092
Description: Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma Pharmacokinetics (PK) parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
  Rac (AUC) is calculated from the ratio of AUC0-tau (Day 15) to AUC0-tau(Day 1).
Time Frame: Day 1：Before administration (within 60 minutes), 0.5, 1, 2, 3, 4, 6, 8, 10 and 12 hours after administration. Day 15: Before administration (within 60 minutes), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours after administration
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | TNP-2092 Capsules 100 mg | TNP-2092 Capsules 300 mg | TNP-2092 Capsules 600 mg
Number analyzed (Participants) | 12 | 12 | 8
ratio | 1.65 (0.54) | 1.51 (0.99) | 1.19 (0.61)

13. Primary Outcome: Accumulation Index Rac(Cmax) of TNP-2092
Description: Plasma concentrations of TNP-2092 were measured by a specific and validated assay. Plasma Pharmacokinetics (PK) parameters of TNP-2092 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods.
  Rac (Cmax) is calculated from the ratio of Cmax (Day 15) to Cmax (Day 1).
Time Frame: as for outcome 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | TNP-2092 Capsules 100 mg | TNP-2092 Capsules 300 mg | TNP-2092 Capsules 600 mg
Number analyzed (Participants) | 12 | 12 | 8
ratio | 1.36 (0.46) | 1.61 (1.56) | 1.24 (0.66)

ADVERSE EVENTS:
Time Frame: Day 1 to Day 49
Description: An Adverse Event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. Preexisting conditions which worsen during a study are also considered as Adverse Events.
Arm/Group | TNP-2092 Capsules 100 mg | TNP-2092 Capsules 300 mg | TNP-2092 Capsules 600 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 6/12 | 9/12 | 4/8 | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TNP-2092 Capsules 100 mg (N=12) | TNP-2092 Capsules 300 mg (N=12) | TNP-2092 Capsules 600 mg (N=8) | Placebo (N=8)
Alanine aminotransferase increased (Investigations) | 3 (5) | 3 (6) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 2 (4) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 2 (2) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Occult blood (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT06190340/Prot_SAP_000.pdf